CLINICAL TRIAL: NCT03129269
Title: Cognitive Function and Prevalence of Amyloid Marker in Frail Older Adults
Acronym: COGFRAIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: MSDAVENIR (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/16/8753
Record Dates: First submitted 2017-03-02; First posted 2017-04-26 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Frail Elderly
Keywords: Cognitive decline; frailty; mild cognitive impairment; Positron Emission Tomography, PET; Alzheimer disease; amyloid load; Magnetic resonance imaging, MRI
MeSH Terms: conditions — Cognitive Dysfunction; Frailty; Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neuroimaging amyloid diagnosis by MRI and PET scan (Experimental): There is only one arm. The procedure consists in neuroimaging to diagnose the presence of amyloid plaques in the brains and permit earlier detection of Alzheimer's disease. MRI and PET Scan.
  * Visits at baseline, 1 and 2 years for a full neuropsychological, functional and physical evaluation.
  * At 6 and 18 months in consultation by a Geriatrician and research assistant for a medical check.
  * one PET-Scan in the 2 months following inclusion for amyloid measurements and one MRI, depending on the clinical relevance
  * A blood sample for biobank at visit 2 and at visit 5.
  Extension study (CogFrail-Plus): additional 2 years follow-up of the COGFRAIL study participants, following the initial 2 years period of the study:
  * 2 Visits at at 36 and 48 months for a full neuropsychological, functional and physical evaluation
  * At 30 and 42 months in consultation by a Geriatrician and research assistant for a medical check
  * A blood sample at 36 and 48 months.
  Interventions: Procedure: MRI and PET scan

INTERVENTIONS:
Procedure: MRI and PET scan — Neuroimaging with MRI and PET scan Amyloid tracer : For PET-scans, 4 MBq/kg of [18F]AV-45 will be injected into each subject in an intravenous bolus.

SUMMARY:
The current study seeks to examine the prevalence of amyloid pathology, among patients referred to the Toulouse Geriatric Frailty Clinic presenting objective memory impairment. We also aim to fully characterize the clinical progression of frail cognitively impaired patients presenting AD (Alzheimer Disease) pathology vs those who also present a cognitive impairment but do not have AD pathology.

DETAILED DESCRIPTION:
The COGFRAIL study is a monocentric study integrating the longitudinal follow-up of 345 individuals referred to the Toulouse Frailty Clinic during 2 years. The procedure consists in neuroimaging to diagnose the presence of amyloid plaques in the brains and permit earlier detection of Alzheimer's disease.

* Visits will be scheduled at baseline, 1 and 2 years for a full neuropsychological, functional and physical evaluation.
* At 6 and 18 months patients will be seen in consultation by a Geriatrician and research assistant for a medical check.
* PET-Scan will be scheduled in the 2 months following inclusion for amyloid measurements. The MRI will be proposed, depending on the clinical relevance
* A blood sample for biobank will be taken at visit 2 and at the end of the study

Extension study (CogFrail-Plus):

The extension study will integrate an additional 2 years follow-up of the

COGFRAIL study participants, following the initial 2 years period of the study:

* 2 Visits will be scheduled at 36 and 48 months for a full neuropsychological, functional and physical evaluation
* At 30 and 42 months patients will be seen in consultation by a Geriatrician and research assistant for a medical check
* A blood sample will be taken at 36 and 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Female and male individuals referred to the Toulouse Frailty Clinic with an objective memory impairment (CDR=0.5 or CDR=1)
* Age ≥ 70 years
* At least 1 Fried-criterion
* Informed consent signed by the patient
* Having an informant accompanying or available by phone
* Individuals affiliated to a healthcare scheme.
* - Willing to be informed in case of a new pathology discovered through medical examination

Extension study (Cog-Frail Plus):

* COGFRAIL study participants still included in the study and completing their last visit (M 24)
* Having a family member or legal representant to sign the consent form if MMSE score <20 at the last visit (M24)

Exclusion Criteria:

* Individuals presenting severe visual or auditory difficulties which may interfere with the completion of neuropsychological and functional assessments.
* Presence of any pathology or severe clinical or psychological condition that, according to the investigator, might interfere with study results or may expose the participants to additional risks.
* Individuals who are robust according to the Fried criteria (0 criteria)
* Individuals who are dependent (Activities of Daily Living (ADL) <4)
* Individuals who have a major deterioration in global cognitive function (Mini Mental State Examination (MMSE) <20)
* Subjects deprived of their liberty by administrative or judicial decision, or under guardianship or admitted to a healthcare or social institution (subjects in non-assisted living facilities could be recruited);

Exclusion criteria for MRI scanning :

* Claustrophobia
* Trauma or surgery which may have left ferromagnetic material in the body, including pacemakers
* History of neurosurgery or aneurism

Extension study (Cog-Frail Plus):

* Presence of any severe pathology that, according to the investigator, might interfere with study results or may expose the participants to additional risks.
* Subjects deprived of their liberty by administrative or judicial decision, or under guardianship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amyloid physiological parameter | 2 months after inclusion
  Amyloid pathology as corroborated with amyloid Positron Emission Tomography (PET) or lumbar punction

SECONDARY OUTCOMES:
Change in cognitive function with Clinical Dementia Rating Scale (CDR) | 12 and 24 months
  Comparison between 2 timeframe to observe change in cognitive function between T12, T24 months
Changes in functional capacities with scales IADL | 12 and 24 months
  Changes in functional capacities, body composition, frailty phenotype, dietary intake and nutritional status with Instrumental Activities of Daily Living (IADL), Activities of Daily Living (ADL), Short Physical Performance Battery (SPPB).
  All measures analysed together, parameters are linked and must be evaluated all together to get the main information.
Changes in functional capacities with scales ADL | 12 and 24 months
  Changes in functional capacities, body composition, frailty phenotype, dietary intake and nutritional status with Instrumental Activities of Daily Living (IADL), Activities of Daily Living (ADL), Short Physical Performance Battery (SPPB).
  All measures analysed together, parameters are linked and must be evaluated all together to get the main information.
Changes in functional capacities with scales SPPB | 12 and 24 months
  Changes in functional capacities, body composition, frailty phenotype, dietary intake and nutritional status with Instrumental Activities of Daily Living (IADL), Activities of Daily Living (ADL), Short Physical Performance Battery (SPPB).
  All measures analysed together, parameters are linked and must be evaluated all together to get the main information.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno VELLAS, MD, Ph D, Pr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robertson DA, Savva GM, Kenny RA. Frailty and cognitive impairment--a review of the evidence and causal mechanisms. Ageing Res Rev. 2013 Sep;12(4):840-51. doi: 10.1016/j.arr.2013.06.004. Epub 2013 Jul 4. PMID 23831959
- [Background] Panza F, Solfrizzi V, Barulli MR, Santamato A, Seripa D, Pilotto A, Logroscino G. Cognitive Frailty: A Systematic Review of Epidemiological and Neurobiological Evidence of an Age-Related Clinical Condition. Rejuvenation Res. 2015 Oct;18(5):389-412. doi: 10.1089/rej.2014.1637. Epub 2015 Aug 20. PMID 25808052
- [Background] Kojima G, Taniguchi Y, Iliffe S, Walters K. Frailty as a Predictor of Alzheimer Disease, Vascular Dementia, and All Dementia Among Community-Dwelling Older People: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2016 Oct 1;17(10):881-8. doi: 10.1016/j.jamda.2016.05.013. Epub 2016 Jun 17. PMID 27324809
- [Background] Buchman AS, Schneider JA, Leurgans S, Bennett DA. Physical frailty in older persons is associated with Alzheimer disease pathology. Neurology. 2008 Aug 12;71(7):499-504. doi: 10.1212/01.wnl.0000324864.81179.6a. PMID 18695161
- [Background] Buchman AS, Yu L, Wilson RS, Schneider JA, Bennett DA. Association of brain pathology with the progression of frailty in older adults. Neurology. 2013 May 28;80(22):2055-61. doi: 10.1212/WNL.0b013e318294b462. Epub 2013 May 1. PMID 23635961
- [Background] Tavassoli N, Guyonnet S, Abellan Van Kan G, Sourdet S, Krams T, Soto ME, Subra J, Chicoulaa B, Ghisolfi A, Balardy L, Cestac P, Rolland Y, Andrieu S, Nourhashemi F, Oustric S, Cesari M, Vellas B; Geriatric Frailty Clinic (G.F.C) for Assessment of Frailty and Prevention of Disability Team. Description of 1,108 older patients referred by their physician to the "Geriatric Frailty Clinic (G.F.C) for Assessment of Frailty and Prevention of Disability" at the gerontopole. J Nutr Health Aging. 2014 May;18(5):457-64. doi: 10.1007/s12603-014-0462-z. PMID 24886728
- [Result] Grande de Franca NA, Diaz G, Lengele L, Soriano G, Caspar-Bauguil S, Saint-Aubert L, Payoux P, Rouch L, Vellas B, de Souto Barreto P, Sourdet S. Associations Between Blood Nutritional Biomarkers and Cerebral Amyloid-beta: Insights From the COGFRAIL Cohort Study. J Gerontol A Biol Sci Med Sci. 2024 Jan 1;79(1):glad248. doi: 10.1093/gerona/glad248. PMID 37879623
- [Result] Sourdet S, Soriano G, Delrieu J, Steinmeyer Z, Guyonnet S, Saint-Aubert L, Payoux P, Ousset PJ, Ghisolfi A, Chicoulaa B, Dardenne S, Gemar T, Baziard M, Guerville F, Andrieu S, Vellas B. Cognitive Function and Amyloid Marker in Frail Older Adults: The COGFRAIL Cohort Study. J Frailty Aging. 2021;10(2):160-167. doi: 10.14283/jfa.2020.57. PMID 33575706
- [Result] Lengele L, Sourdet S, Soriano G, Rolland Y, Soler V, de Souto Barreto P. Cross-sectional associations of dietary intake with hearing and vision capacities and potential mediation effect of inflammation in older adults: the COGFRAIL study. Aging Clin Exp Res. 2023 Jun;35(6):1325-1337. doi: 10.1007/s40520-023-02418-7. Epub 2023 Apr 29. PMID 37119508
- [Derived] Bellelli F, Delrieu J, van Kan GA, Peluso A, Soriano G, Vellas B, Angioni D, Sourdet S. Are pre-frail and frail amyloid positive individuals eligible to Lecanemab? A cross-sectional analysis from the Cogfrail real-world cohort. Alzheimers Res Ther. 2026 Feb 4. doi: 10.1186/s13195-026-01966-0. Online ahead of print. PMID 41634843